CLINICAL TRIAL: NCT04257903
Title: Effectiveness of Different Treatment Methods in Patients With Myofascial Pain Syndrome
Brief Title: Different Treatment Modalities for Myofascial Pain
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Aysegul Kurt, Assistant Professor, Trakya University
Other Study IDs: TUFT-BAEK 2019/114
Record Dates: First submitted 2020-01-28; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Myofascial Pain; Splints; Low-Level Laser Therapy
Keywords: Myofacial Pain; Occlusal Splint; Low-Level Laser Therapy
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Occlusal Splint Therapy: The data of patients who previously received occlusal splint therapy were evaluated. Participants in the study received occlusal splint therapy, but the investigator did not assign this intervention specifically to the study participants. Participants received occlusal splint therapy as part of routine medical care, and a researcher studied the effect of occlusal splint therapy.
- Low-Level Laser Therapy: The data of patients who previously received Low-Level Laser Therapy were evaluated. Participants in the study received Low-Level Laser Therapy, but the investigator did not assign this intervention specifically to the study participants. Participants received Low-Level Laser Therapy as part of routine medical care, and a researcher studied the effect of Low-Level Laser Therapy.

SUMMARY:
Myofascial pain dysfunction syndrome (MPDS) is the most common reason for pain and limited function of the masticatory system. The low-level laser therapy (LLLT) and occlusal splint therapy (OST) are therapeutic options for MPDS. This study aims to evaluate the effect of LLLT and OST on pain relief and mandibular movement improvement in patients with myofascial pain.

DETAILED DESCRIPTION:
Myofascial pain dysfunction syndrome in the masticatory muscles is the most common temporomandibular disorder. Patients suffer from pain and muscle tenderness and may present with or without restricted mouth opening. The etiology of myofascial pain dysfunction syndrome is multifactorial including psychological factors, occlusion imbalance, and parafunctional habits. Treatments for myofascial pain dysfunction syndrome include education, self-care, physical therapy, use of intra-oral appliances, short-term pharmacotherapy, behavioral therapy, and relaxation techniques.

Temporomandibular disorder is most often treated using occlusal splints safely to reduce temporomandibular joint load, and subsequently, clinical symptoms, as a reversible therapy. Occlusal splints need to be used for at least three months to eliminate temporomandibular disorders.

One of physical therapy is laser treatment. Laser treatment on tissues provides a clinical effect called biostimulation, where the basic mechanism occurs at the molecular level.

The low-level laser has non-invasive and inoffensive characteristics at appropriate parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myofascial pain syndrome according to The Research Diagnostic Criteria for Temporomandibular Disorder.
* Individuals between the ages of 18-60
* Occlusion of individuals with posterior teeth
* Forms of individuals who do not have any systemic disease

Exclusion Criteria:

* Disc displacement with or without reduction, with or without limited mouth opening, arthralgia, arthritis, arthrosis
* Inflammatory connective tissue disease (such as rheumatoid arthritis)
* Psychiatric diseases
* Tumor
* Heart diseases
* Pregnancy
* Diseases that may cause pain symptoms in other orofacial regions (toothache, neuralgia, migraine)
* Having received any treatment for headache or bruxism in the last 2 years
* Skin infections on the masseter and temporal muscles

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Thracian region
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Visual Analogue Scale | Baseline, one month after the beginning of treatment and two months after the beginning of treatment
  Pain intensity during muscle palpations. Scores are ranging from 0 to 10. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change from Baseline maximum unassisted mouth opening | Baseline, one month after the beginning of treatment and two months after the beginning of treatment
  Value of Maximum unassisted mouth opening as a centimeter. Scores are ranging from 0 to 45 centimeters. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Merkez, Edirne, Turkey (Türkiye)